CLINICAL TRIAL: NCT02929524
Title: Intranasal Ketamine for Peripheral Venous Puncture in Pediatric Patients: A Randomized Double Blind and Placebo Controlled Study
Brief Title: Intranasal Ketamine as a Sedative for Venipuncture
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 150424
Record Dates: First submitted 2016-10-07; First posted 2016-10-11 (Estimated); Last update posted 2016-10-11 (Estimated); Status verified 2016-10

CONDITIONS: Respiratory Tract Disease; Acute Pain; Diseases of the Digestive System
Keywords: Ketamine; Intranasal administration; Pediatric nursing
MeSH Terms: conditions — Respiratory Tract Diseases; Acute Pain; Digestive System Diseases | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine group (Experimental): This group was used intranasal ketamine, syringes were made with 4 ml of the drug (50mg/ml), 1 randomized per patient. The validity stability and were 7 days after drawing the solution. The drug began to take effect in 10 minutes and lasted about 40 minutes.
  Interventions: Drug: Ketamine
- Placebo Group (Placebo Comparator): This group was used intranasal saline, syringes were made with 4 ml of liquid 1 per patient randomized. The validity stability and were 7 days after drawing the solution.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine — As indicated the use of sedative and after authorization of the person responsible, the child receives the intranasal solution. Before administration of the solution 2 hour and 24 hours after the procedure, must be recorded vital signs of the patient. A person with the help of a clock will make the time count. The nurse and the patient's family must respond to the study protocol questions
  Other Names: Intervention group
  Arms: Ketamine group
Drug: Placebo — As indicated the use of sedative and after authorization of the person responsible, the child receives the intranasal solution. Before administration of the solution 2 hour and 24 hours after the procedure, must be recorded vital signs of the patient. A person with the help of a clock will make the time count. The nurse and the patient's family must respond to the study protocol questions
  Other Names: Saline group
  Arms: Placebo Group

SUMMARY:
Randomized clinical trial, controlled, double-blind, parallel two-arm.

DETAILED DESCRIPTION:
Randomized, double-blind, placebo controlled study conducted at the Clinical Hospital of Porto Alegre between November / 15 and August / 16. This study was approved by the Ethics Committee of the Institution. Participated children requiring venipuncture randomized in the intervention group who received the ketamine IN 4 mg/kg and placebo saline group. The groups were compared: Puncture time, ease the nurse to perform the procedure, adverse events, changes in vital signs and perception of the companion.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized in the Pediatric Inpatient Units, with the presence of legal guardian;
* Aged 3 months to 12 years;
* Requiring venipuncture independent research.

Exclusion Criteria:

* Severe neurological sequelae;
* Patients who need immediate venipuncture at risk;
* Presence of active nosebleeds;
* Patients using drugs sedative and analgesic continuos;
* Children who have experienced clinical change with ketamine.

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2015-04; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Decreased venipuncture Time | Expected 3 minutes difference between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson Piva, Study Director — Hospital de Clinicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided